CLINICAL TRIAL: NCT03384836
Title: A Phase Ib/II Study of Propranolol With Fixed-Dose Pembrolizumab in Patients With Unresectable Stage III and Stage IV Melanoma
Brief Title: Propranolol Hydrochloride and Pembrolizumab in Treating Patients With Stage IIIC-IV Melanoma That Cannot Be Removed by Surgery
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: interim Analysis
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 53217; NCI-2017-02210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 53217 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2017-12-12; First posted 2017-12-27 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
Keywords: Melanoma; Immune Checkpoint Inhibitors; Beta Adrenergic Blockers
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Propranolol; propranolol CR

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (propranolol hydrochloride, pembrolizumab) (Experimental): Patients receive propranolol hydrochloride PO BID and pembrolizumab IV over 30 minutes of day 1. Courses repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Drug: Propranolol Hydrochloride

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Propranolol Hydrochloride — Given PO
  Other Names: Inderal; Innopran XL

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of propranolol hydrochloride when given together with pembrolizumab and how well they work in treating patients with stage IIIC-IV melanoma that cannot be removed by surgery. Pembrolizumab is a monoclonal antibody that "takes the brakes off the immune system" and thus allows for anti-tumor immune responses. Propranolol hydrochloride is a beta adrenergic blocking agent that can enhance immune cell responses when under stress. Giving propranolol hydrochloride and pembrolizumab may work better in treating patients with melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine dose limiting toxicities (DLT) of propranolol hydrochloride (propranolol) in combination with fixed dose pembrolizumab in the treatment of melanoma.

II. To evaluate the efficacy of pembrolizumab in combination with propranolol in patients with melanoma, as determined by overall response rate (ORR) per immune-modified Response Evaluation Criteria in Solid Tumors (RECIST) (1).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of pembrolizumab in combination with propranolol in patients with melanoma, as determined by secondary measures of efficacy, including: progression free survival (PFS) and overall survival (OS).

TERTIARY OBJECTIVES:

I. To correlate baseline or changes in the levels of biomarkers, like, peripheral T-cell subsets/myeloid derived suppressor cells (MDSC)/cytokines/urinary catecholamine and perceived stress scale (PSS) with efficacy (ORR, PFS, OS) in melanoma patients treated with pembrolizumab and propranolol.

OUTLINE: This is a phase Ib, dose-escalation study of propranolol hydrochloride followed by a phase II study.

Patients receive propranolol hydrochloride orally (PO) twice daily (BID) and pembrolizumab intravenously (IV) over 30 minutes of day 1. Courses repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 6 months, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be newly diagnosed, treatment-naive with histologically confirmed stage IIIC unresectable melanoma or stage IV melanoma
* Have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Available archival formalin-fixed paraffin-embedded (FFPE) from a prior biopsy or, participant must be willing to have a tissue biopsy taken at a clinic visit prior to start of study treatment
* Have measurable disease per irRECIST v1.1
* Ability to swallow and retain oral medication
* Absolute neutrophil count (ANC) >= 1500/uL
* Hemoglobin (Hb) >= 9 g/dL
* Platelet count >= 100, 000/uL
* Total bilirubin =< 1.5 x ULN (upper limit of normal) - unless patient has Gilbert's syndrome
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2 x ULN
* If the patient has liver metastasis AST and ALT less than or greater to 5x ULN
* Serum or plasma (based on site's SOP) creatinine < 2 x ULN
* Participants of child-bearing potential must have a negative pregnancy test at study entry and then agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Participants who have received previous immunotherapy for any cancer (excluding melanoma) including PD-1/PD-L1 inhibitors but not interferons and CTLA-4 inhibitors
* Participants with chronic autoimmune diseases
* Participants that are already on non-selective B-AR blockers for various indications. Patients on selective beta-blockers are considered eligible for enrollment with a caveat that their clinician prescribing the beta-blocker is willing to discontinue their selective beta-blocker in order to transition to propranolol at the specified protocol dose.
* Participants with symptomatic known brain metastases < 4 weeks from radiation treatment should be excluded from this clinical trial
* Other invasive cancers diagnosed < 3 years back that required systemic treatment. If diagnosed with other invasive cancer >=3 years, should have complete recovery from all systemic toxicity except neuropathy and alopecia
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female participants, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Other active non-melanoma metastatic cancers
* Contraindications to the use of beta-blockers, like, uncontrolled depression, unstable angina pectoris, uncontrolled heart failure (grade III or IV), hypotension (systolic blood pressure < 100 mmHg), bradycardia (resting heart rate <55bpm), severe asthma or chronic obstructive pulmonary disease (COPD), uncontrolled type I or type II diabetes mellitus (glycosylated hemoglobin [HbA1C] > 8.5 or fasting plasma glucose > 160 mg/dl at screening), symptomatic peripheral arterial disease or Raynaud's syndrome, untreated pheochromocytoma, current use or past use in the last two years of non-selective beta-blockers or non-dihydropyridine calcium channel blockers. Patients on selective beta blockers will be eligible for enrollment only under the condition that their prescribing clinician is willing to discontinue their selective beta blocker in order to begin propranolol and only at the specified dose (after which time the patient is not to be started on any non-selective beta-blockers or non-dihydropyridine calcium channel blockers)
* Patient is currently receiving or has received systemic corticosteroids (=< 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment)
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of the study drug
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) defined as any grade 3 or higher hematological or non-hematological toxicity that is probably or definitely related to treatment according to Common Terminology Criteria for Adverse Events version 4.03 (Phase Ib) | Up to 12 weeks
  Adverse events and toxicities will be summarized by dose level using frequencies and relative frequencies.
Overall response rate (ORR) per immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) version 1.1 (Phase II) | Up to 6 months
  ORR is defined as partial or complete response within 6 months of initiating combination therapy.

SECONDARY OUTCOMES:
Overall survival (OS) (Phase II) | From treatment initiation until death due to any cause (event) or last follow-up, assessed up to 2 years
  Will be summarized using standard Kaplan-Meier methods and rates will be obtained with 90% confidence intervals.
PFS (Phase II) | From treatment initiation until disease progression, death due to disease (events), or last follow-up, assessed up to 2 years
  Will summarized using standard Kaplan-Meier methods and rates will be obtained with 90% confidence intervals.
Progression free survival (PFS) (Phase II) | At 1 year
  Will be summarized using standard Kaplan-Meier methods and rates will be obtained with 90% confidence intervals.

OTHER OUTCOMES:
Changes in the levels of biomarkers | Baseline up to 2 years
  to correlate baseline or changes in levels of biomarkers with efficacy in melanoma patients treated with pembrolizumab and propranolol.

CONTACTS AND LOCATIONS:
Overall Officials: Shipra Gandhi, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (4):
- United States (4):
  - Emory University Hospital/ Winship Cancer Institute, Atlanta, Georgia
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Penn State Milton S. Hershy Medical Center Cancer Institute, Hershey, Pennsylvania